CLINICAL TRIAL: NCT05480501
Title: Clinical Trial to Evaluate the Safety and Efficacy of IM19 CAR-T Cells in Patients With Relapsed and Refractory (R/R) B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART1902
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Leukemia
Keywords: CAR-T; B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia; Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CAR-T cells (Experimental)
  Interventions: Biological: IM19 CAR-T cells

INTERVENTIONS:
Biological: IM19 CAR-T cells — IM19 CAR-T cells administrated in a dosage to be selected by physician from a specific range.

SUMMARY:
This is a open-label to assess the efficacy and safety of IM19 CAR-T cells in R/R B-cell Acute Lymphoblastic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-ALL, defined as：1）Not chieving a CR after 1 cycle of standard chemotherapy for relapsed leukemia. 2）Any relapse after HSCT and must be ≥ 6 months from HSCT at the time of IM19 CAR-T cells infusion. 3）Primary refractory as defined by not achieving a CR after 2 cycles of a standard chemotherapy regimen.
* Patients with Ph+ ALL are eligible if they are intolerant to or have failed two lines of TKI ± chemotherapy ；Ph + all patients with T315I mutation are not required to receive at least two TKI ± chemotherapy in the absence of effective TKI therapy.
* Morphological evidence of disease in bone marrow (at least 5% blasts).
* Aged 3 to 70 years.
* Estimated life expectancy >3 months.
* ECOG performance status of 0 or 1(age ≥ 16 years) or Lansky (age < 16 years).
* Women of childbearing age who had a negative blood pregnancy test before the start of the trial and agreed to take effective contraceptive measures during the trial period until the last follow-up; male subjects with fertility partners agreed to take effective contraceptive measures during the trial period until the last follow-up.
* Adequate organ function.
* Volunteer to participate in this trial and sign on the informed consent.

Exclusion Criteria:

* Subjects with lsolated extramedullary disease relapse.
* Subjects with Burkitt's lymphoma.
* Subjects has obvious symptoms of central nervous system invasion and needs targeted treatment.
* Subjects has previously received gene product therapy.
* Subjects has graft-versus-host response（GVHD） and need to use immunosuppressants or GVHD ≥ grade 2 or being treated with anti GVHD or suffering from autoimmune diseases.
* Subjects has received chemotherapy or radiotherapy within 3 days before leukapheresis.
* Subjects received systemic steroids within 5 days prior to leukapheresis.
* Subjects received drugs that stimulated the production of hematopoietic cells in the bone marrow for 5 days prior to leucapheresis.
* Subjects has participated in other clinical studies within 1 month before screening or plan to participate in other drug clinical trials during this study.
* Subjects received allogeneic cell therapy within 6 weeks before leukapheresis.
* Subjects with History or presence of CNS disorder.
* Subjects with HBV, HCV, HIV ,EBV,ECV or syphilis infection at the time of screening.
* Pregnant or lactating, or planning pregnancy within 180 days after the end of CAR-T cells infusion, or male patients whose partners plan pregnancy 180 days after their CAR-T cell infusion.
* Subjects with other tumors in the past 5 years.
* Within 14 days before enrollment, there were active or uncontrollable infections requiring systemic treatment.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 28 days after CAR-T cell infusion
Persistence of CAR-T cells (cell counts and cell percentage in peripheral blood and bone marrow ) | Up to 24 weeks after CAR-T cell infusion

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 weeks after CAR-T cell infusion
Relapse free surviva（PFS） | Up to 24 weeks after CAR-T cell infusion
Duration of Response (DOR) | Up to 24 weeks after CAR-T cell infusion
Overall survival (OS) | Up to 24 weeks after CAR-T cell infusion
Minimal residual disease（MRD） | Up to 24 weeks after CAR-T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Yan, M.D., Principal Investigator — Hospital of China Medical University
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China